CLINICAL TRIAL: NCT01348373
Title: Evaluation of Effectiveness and Safety of the GENOUS STENT in ST-Segment Elevation Myocardial Infarction
Brief Title: Evaluation of Effectiveness and Safety of the GENOUS STENT (IRIS-GENOUS STEMI)
Status: Completed | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other); OrbusNeich Medical Korea Co., Ltd. (Unknown)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, Chairman,Heart Institute, Asan Medical Center,University of Ulsan,College of Medicine, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Other Study IDs: CVRF2010-05
Record Dates: First submitted 2011-05-04; First posted 2011-05-05 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Coronary Artery Disease
Keywords: drug eluting stents
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- GENOUS EPC-coated stent: Patients treated with GENOUS EPC-coated stent

SUMMARY:
The objective of this study is to evaluate effectiveness and safety of GENOUS EPC-coated stent in patients with STEMI with other drug-eluting stents (DESs).

DETAILED DESCRIPTION:
This study is a non-randomized, prospective, open-label registry to compare the efficacy and safety of GENOUS stent in STEMI patients with other-type DESs.

ELIGIBILITY:
Inclusion Criteria:

* STEMI Patients requiring primary PCI.
* The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethics Committee of the respective clinical site

Exclusion Criteria:

* Patients with a mixture of other DESs
* Terminal illness with life expectancy <1 year
* Patients with cardiogenic shock

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: STEMI Patients requiring primary PCI.
Sampling Method: Non-Probability Sample
Enrollment: 464 (Actual)
Dates: Start 2010-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
composite of death, nonfatal myocardial infarction (MI), or ischemic-driven Target- Vessel Revascularization (TVR) | 12 months post procedure

SECONDARY OUTCOMES:
Death (all cause and cardiac) | one month
Death (all cause and cardiac) | 6 months
Death (all cause and cardiac) | yearly up to 5 years
MI | one month
MI | 6 months
MI | yearly up to 5 years
Composite of death or MI | one month
Composite of death or MI | 6 months
Composite of death or MI | yearly up to 5 years
Composite of cardiac death or MI | one month
Composite of cardiac death or MI | 6 months
Composite of cardiac death or MI | yearly up to 5 years
TVR | one month
TVR | 6 months
TVR | yearly up to 5 years
Target-lesion revascularization (TLR) | yearly up to 5 years
Target-lesion revascularization (TLR) | one month
Target-lesion revascularization (TLR) | 6 months
Stent thrombosis (ARC criteria) | one month
Stent thrombosis (ARC criteria) | 6 months
Stent thrombosis (ARC criteria) | yearly up to 5 years
Procedural success (defined as achievement of a final diameter stenosis of <30% by visual estimation, without the occurrence of death, Q-wave MI, or urgent revascularization during the index hospitalization) | in-hospital

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, PhD, Principal Investigator — Asan Medical Center; Ki Bae Seung, MD, PhD, Principal Investigator — Seoul St. Mary's Hospital, Catholic University of Korea
Locations (16):
- South Korea (16):
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Kangwon National University Hospital, Chuncheon
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Konyang University Hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Chonnam National University Hospital, Gwangju
  - National Health Insurance Corporation Ilsan Hospital, Ilsan
  - Gachon University Gil Hospital, Incheon
  - Inha University Hospital, Incheon
  - Pusan National University Yangsan Hospital, Pusan
  - Asan Medical Center, Seoul
  - Kangbuk Samsung Medical Center, Seoul
  - SMA-SNU Boramae Medical Center, Seoul
  - Ulsan University Hospital, Ulsan
  - Wonju Christian Hospital, Wŏnju